CLINICAL TRIAL: NCT06179550
Title: A Randomized Controlled Study to Explore the Clinical Effect of Intermittent Oro-esophageal Tube Feeding vs. Nasogastric Tube Feeding on Cerebral Small Vessel Disease Patients With Dysphagia
Brief Title: Intermittent Oro-esophageal Tube Feeding on Cerebral Small Vessel Disease Patients With Dysphagia
Acronym: CSVD
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: ethical issues
Sponsor: Zeng Changhao (Other)
Responsible Party: Sponsor-Investigator, Zeng Changhao, PI, People's Hospital of Zhengzhou University
Organization: People's Hospital of Zhengzhou University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2022-KY-1532; Zhengzhou University (Registry Identifier: kfkioecsvd)
Record Dates: First submitted 2023-12-02; First posted 2023-12-22 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Cerebral Small Vessel Diseases
Keywords: Cerebral Small Vessel Disease; Enteral Nutrition.; Intermittent Oro-esophageal Tube Feeding
MeSH Terms: conditions — Cerebral Small Vessel Diseases | interventions — Enteral Nutrition

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: The researchers respectively responsible for intervention, assessment, and data collection maintained an isolated status from the patients enrolled beyond the necessary contact, strictly adhering to the principle of not disclosing group information. Furthermore, the trained professionals who were not involved in the intervention were selected to conduct all assessments, data collection, and analysis to ensure the objectivity and independence of result evaluation. All medical personnel involved in interventions received detailed training to ensure their understanding and proper implementation of the interventions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The control group (Active Comparator): Assigned by the random number table. During the treatment, all patients were provided with comprehensive rehabilitation therapy as follows:
  1. Basic treatment, including corresponding control of risk factors and education on healthy lifestyles.
  2. Swallowing training, including lemon ice stimulation, mendelson maneuver, empty swallowing training, and pronunciation training.
  3. Pulmonary function training, including standing training, cough training, and diaphragm muscle training.
  Besides, the control group was given enteral nutritional support with NGT according to the relevant guidelines. Within 4 hours after admission, the placement of the feeding tube was conducted by professional medical staffs and after intubation, the tube was secured to the patient's cheek with medical tape. The feeding was conducted once every 3-4 hours, with 200-300ml each time. The total feeding volume was determined based on daily requirements.
  Interventions: Device: Nasogastric tube
- The observation group (Experimental): Assigned by the random number table.During the treatment, all patients were provided with comprehensive rehabilitation therapy as follows:
  1. Basic treatment, including corresponding control of risk factors and education on healthy lifestyles.
  2. Swallowing training, including lemon ice stimulation, mendelson maneuver, empty swallowing training, and pronunciation training.
  3. Pulmonary function training, including standing training, cough training, and diaphragm muscle training.
  The observation group was given enteral nutritional support with IOE according to the following procedure. The feeding content was formulated by the nutritionists based on the patient's condition and relevant guidelines to reach the energy demand as 20-25 kcal/kg/day and protein supplementation of 1.2-2.0 g/kg/day for both two groups
  Interventions: Device: Intermittent Oro-esophageal Tube

INTERVENTIONS:
Device: Nasogastric tube — Besides, the control group was given enteral nutritional support with NGT according to the relevant guidelines. Within 4 hours after admission, the placement of the feeding tube was conducted by professional medical staffs and after intubation, the tube was secured to the patient's cheek with medical tape. The feeding was conducted once every 3-4 hours, with 200-300ml each time. The total feeding volume was determined based on daily requirements. The feeding content was formulated by the nutritionists based on the patient's condition and relevant guidelines to reach the energy demand as 20-25 kcal/kg/day and protein supplementation of 1.2-2.0 g/kg/day for both two groups. For patients with limited tube feeding compliance, we made appropriate adjustments to ensure that they were not at risk of severe malnutrition as much as possible.
  Other Names: 1) Basic treatment, including corresponding control of risk factors and education on healthy lifestyles.; 2) Swallowing training, including lemon ice stimulation, mendelson maneuver, empty swallowing training, and pronunciation training.; 3) Pulmonary function training, including standing training, cough training, and diaphragm muscle training.
  Arms: The control group
Device: Intermittent Oro-esophageal Tube — The observation group was given enteral nutritional support with IOE according to the following procedure: Before each feeding, inside and outside of the tube was cleaned with water. During feeding, the patient should maintain a semi-reclining or sitting position with mouth opened, and the tube was inserted slowly and smoothly into the upper part of the esophagus by medical staffs while the appropriate depth of intubation was checked with the calibration markings on the tube wall. The distance from the incisors to the head part of the tube should be between 22-25 cm (Appendix). However, the specific depth should be evaluated based on patients' feedback and adjusted accordingly. After insertion, the tail part of the tube should be put into a container full of water and the absence of continuous bubbles indicated a successful intubation. Then, the feeding was to be conducted three times per day with 50 ml per minute and 400-600ml for each feeding.
  Other Names: 1) Basic treatment, including corresponding control of risk factors and education on healthy lifestyles.; 2) Swallowing training, including lemon ice stimulation, mendelson maneuver, empty swallowing training, and pronunciation training.; 3) Pulmonary function training, including standing training, cough training, and diaphragm muscle training.
  Arms: The observation group

SUMMARY:
Nasogastric tube feeding (NGT) has been widely used in cerebral small vessel disease (CSVD) patients with dysphagia but has a significant risk of complications. Intermittent Oro-esophageal Tube Feeding (IOE) is an established enteral nutrition approach that can be used with comprehensive rehabilitation therapy. This study aims to explore the clinical effect of IOE vs. NGT on CSVD Patients with Dysphagia. Compared to NGT, IOE, as an enteral nutrition support mode, in CSVD Patients with Dysphagia who received comprehensive rehabilitation therapy, showed advantages in improvement in dysphagia, nutritional status, ADL, QOL, pneumonia, and adverse events, which should be considered as the preferred approach.

DETAILED DESCRIPTION:
Nasogastric tube feeding (NGT) has been widely used in cerebral small vessel disease (CSVD) patients with dysphagia but has a significant risk of complications. Intermittent Oro-esophageal Tube Feeding (IOE) is an established enteral nutrition approach that can be used with comprehensive rehabilitation therapy. This study aims to explore the clinical effect of IOE vs. NGT on CSVD Patients with Dysphagia.

This was a randomized controlled study with 60 CSVD Patients with Dysphagia who received comprehensive rehabilitation therapy. Patients enrolled were randomly divided into the observation group (with IOE, n=30) and the control group (with NGT, n=30). At admission and after treatment, Video Fluoroscopic Swallowing Study (VFSS) and Functional Oral Intake Scale (FOIS), body mass index (BMI), serum albumin (Alb), and hemoglobin (Hb), Modified Barthel Index (MBI) and World Health Organization Quality of Life Assessment Instrument Brief Version (WHOQOL-BREF) were recruited to assess and compare dysphagia, nutritional status, activities of daily living (ADL) and quality of life (QOL). The incidence of pneumonia was recorded and compared.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of CSVD, confirmed by MRI;
* Must be able to cooperate with treatment and questionnaire investigation, (Generally with a Mini-Mental State Examination (MMSE) score ≥ 24) ;
* Clinical diagnosis of dysphagia through the Functional Oral Intake Scale (FOIS) and Video Fluoroscopic Swallowing Study (VFSS);
* Age between 40 and 70 years;
* Enteral nutrition support was required and feasible.
* No history of prior stroke.

Exclusion Criteria:

* Dysphagia related to other cerebrovascular diseases or caused by neurodegenerative diseases;
* Complicated with severe liver and kidney failure, tumors, or hematological disorders;
* Simultaneously need to undergo other therapy that might affect the outcomes of this study;
* Unable or unwilling to undergo VFSS;
* Pregnant or nursing females.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-06-03 (Actual); Study Completion 2023-06-22 (Actual)

PRIMARY OUTCOMES:
Video Fluoroscopic Swallowing Study | day 1 and day 15
  Video Fluoroscopic Swallowing Study, which is considered as the "gold standard", swallowing process is divided into four periods: cognitive, oral, pharyngeal, and esophageal periods with a total score of 10 and a higher score indicates better swallowing ability (less dysphagia).

SECONDARY OUTCOMES:
Functional Oral Intake Scale | day 1 and day 15
  During Dysphagia-Functional Oral Intake Scale assessment, evaluators engage in communication with the patient, conduct observations, and make records to assess the patient's oral intake ability. The FOIS assessment form includes seven levels of scoring, ranging from level 1 to level 7, indicating a progressive improvement in the patient's oral intake ability. In general, the result below level 6 indicates unsafe for oral intake while level 6 and above indicates that eating via mouth can be safely conducted.
Body mass index | day 1 and day 15
  Weight and height will be combined to report Body mass index in kg/m^2
Serum albumin | day 1 and day 15
  Serum albumin was recorded via blood routine test.(Alb, g/L)
Hemoglobin | day 1 and day 15
  Hemoglobin was recorded via blood routine test.(Hb, mg/L)
Pneumonia | day 1 and day 15
  The occurrence of pneumonia in patients was assessed before and after treatment. Specifically, first of all, the symptom assessment and physical examination were conducted to all patients, during which, the doctor would inquire symptoms related to pneumonia, such as cough, sputum production, difficulty breathing, chest pain, etc. and observe the patient's respiratory condition, including respiratory rate, breath sounds, and any abnormal signs in the chest. If there was probability for potential pneumonia, patients were requested to undergo lung CT for further diagnosis
Activities of daily living | day 1 and day 15
  The activities of daily living was assessed utilizing the Modified Barthel Index (MBI). Modified Barthel Index includes the following 10 subscales. For each subscale, choices encoded with the score 10, 8, 5, 2, 0 are set with the decreasing level of self-dependence, while the final total is positively correlated with Activities of daily living. Cronbach's α of questionnaire adopted is 0.916.
World Health Organization Quality of Life Assessment Instrument Brief Version | day 1 and day 15
  The Quality of Life was assessed utilizing the World Health Organization Quality of Life Assessment Instrument Brief Version (WHOQOL-BREF). WHOQOL-BREF covers various aspects such as mobility, pain, emotions, personal relationships, living conditions, and access to health services, to evaluate Quality of Life. Each item is rated on a Likert scale, and the scores are transformed into a standardized score ranging from 0 to 100, with higher scores indicating better Quality of Life.

CONTACTS AND LOCATIONS:
Overall Officials: Nieto Luis, Master, Principal Investigator — Site Coordinator of United Medical Group located in Miami
Locations (1):
- Zheng da yi fu yuan hospital, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No
The datasets generated and analyzed during the current study are not publicly available due to Data Confidentiality of National Key R&D Projects but are available from the corresponding author on reasonable request.

DOCUMENTS (3):
  • Study Protocol (2022-12-01): https://cdn.clinicaltrials.gov/large-docs/50/NCT06179550/Prot_000.pdf
  • Statistical Analysis Plan (2022-12-10): https://cdn.clinicaltrials.gov/large-docs/50/NCT06179550/SAP_001.pdf
  • Informed Consent Form (2022-12-10): https://cdn.clinicaltrials.gov/large-docs/50/NCT06179550/ICF_002.pdf